CLINICAL TRIAL: NCT03893773
Title: Doppler Ultrasonography in Assessment of Graft Hemodynamics After Living-Donor Liver Transplantation in Al-Rajhi Liver Hospital
Brief Title: Doppler Ultrasonography in Assessment of Graft Hemodynamics After Living-Donor Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ZRMohamed (Other)
Responsible Party: Sponsor-Investigator, ZRMohamed, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: DAGHALDLTAL
Record Dates: First submitted 2019-03-24; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Liver Transplant, Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: doppler ultrasonagraphy — The following parameters will be measured:
  Hepatic artery Resistance index (HARI), Diameter, peak systolic velocity (HAPSV, cm/s).
  Portal vein peak velocity (PVPV) and diameter at the anastomotic and non-anastomotic sites.
  Hepatic vein peak velocity and wave form

SUMMARY:
Graft ischemia after liver transplantation is associated with a high incidence of morbidity and mortality . The overall incidence of vascular complications in adults varies widely among transplant centers worldwide, but remains around 7% in various series of deceased donor liver transplantation (DDLT), and around 13% involving living donor liver transplantation (LDLT) Vascular complications include; hepatic artery thrombosis and stenosis, portal vein thrombosis and stenosis, caval and hepatic veins obstruction, arterial pseudo aneurysm. Biliary complications include; biliary leakage, stricture and obstruction .

DETAILED DESCRIPTION:
Hepatic artery thrombosis (HAT) is the most severe and frequent complication represents more than 50% of all arterial complications. Early HAT occurring within 1 month post-operation in 2.9%, and late HAT in 2.2%. The overall mortality rate for patients with early HAT is about 33% (13).

Hepatic arterial stenosis can occur immediately postoperative or later with an incidence of 1% to 2% and has been suggested to progress to HAT. This is due to surgical technique or fibrotic healing (14).

Hepatic artery aneurysm or pseudoaneurysm is rare and has an incidence of 0.27-3%. They occur in the second or third post-transplant week after infection caused by biliary sepsis, intestinal perforation, anastomotic leak, or intrahepatic stenting, or technical failure .

Portal vein thrombosis (partial or complete) or stenosis has an incidence of 2-3%, it can occur early postoperative within 1 month or more late. Early portal vein thrombosis can lead to liver insufficiency and failure. Late presentation, depending on the collateral circulation, can lead to portal hypertension with varices and ascites .

Currently, transplant outflow obstruction by kinking, stenosis or thrombosis of the inferior vena cava (IVC) or hepatic vein, especially in LDLT, are relatively uncommon complications following liver transplantation with an reported incidence of less than 3%. The main risk factor is a technical error in the creation of the anastomosis Despite all the advances in transplant patient care and surgical techniques, biliary complications remain high incidence in living donor or split liver transplant. There are early and late complications, and there are anastomotic, and nonanastomotic biliary complications, such as stones, sludge and casts .

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 y with living donor liver transplantation in Al-Rajhi liver hospital, Assiut, Egypt

Exclusion Criteria:

* Pediatric liver transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults more than 18 y with living donor liver transplantation in Al-Rajhi liver hospital, Assiut, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of vascular complication: | 6 month after liver transplantation.
  A. Hepatic artery thrombosis (HAT), stenosis (HAS). B. Portal vein thrombosis (PVT), or stenosis. C. Hepatic veins and inferior vena cava thrombosis, or stenosis. The investigator will record nature of the complication, time of presentation and Number of hospital re-admissions (due to vascular complications).
Intervention done due to vascular complication | 6 month after liver transplantation
  Non-surgical intervention (percutaneous transluminal angioplasty (PTA) +/- stent placement, catheter-directed thrombolysis, thrombectomy, trans-catheter arterial embolization) or surgical revision with detailed description of each intervention and if the intervention is successful or not (improvement of symptom and liver function).